CLINICAL TRIAL: NCT03485508
Title: Imaging and Risk Stratification in the Brugada Syndrome: a Follow-up Study
Brief Title: The Brugada Syndrome: a Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/253
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-02

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome | interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Transthoracic echocardiography Blood sample with assessment of biomarkers
  Other Names: Blood sample

SUMMARY:
Although for many years the Brugada syndrome has been labelled as a purely electrical disease in the structurally normal heart, the evolution of imaging techniques has enabled the discovery of subtle morphofunctional alterations in some of the Brugada syndrome patients. We will use new echocardiographic techniques to assess cardiac function in these patients and new parameters will be evaluated for their prognostic value as risk stratificators.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of Brugada syndrome

Exclusion Criteria:

* history of pericarditis, ischemic heart disease, cardiomyopathy of any origin, structural heart disease, or any other channelopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Brugada syndrome patients visiting the UZ Brussel for diagnosis or follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-03-11 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Composed outcome of sudden cardiac death, appropriate ICD shock and witnessed ventricular fibrillation | 6 years
  Sudden cardiac death is death occuring within 24 hours after being seen in a healthy status or within 1 hour after initiation of symptoms.

SECONDARY OUTCOMES:
Syncope | 6 years
  Loss of consciousness

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided